CLINICAL TRIAL: NCT02631824
Title: Radiologic and Clinical Outcomes of Augmentation in Fragility Intertrochanteric Hip Fracture Treatment: A Randomized Multicenter Clinical Trial
Brief Title: Radiologic and Clinical Outcomes of Augmentation in Fragility Intertrochanteric Hip Fracture Treatment
Acronym: AFIF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Infantil Universitario de San Jose (Other)
Collaborators: Fundación Santa Fe de Bogota (Other)
Responsible Party: Principal Investigator, Carlos Mario Olarte, Head of Orthopedics Department at HIUSJ, Hospital Infantil Universitario de San Jose
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HIPFX-001-AUGM
Record Dates: First submitted 2015-12-05; First posted 2015-12-16 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Hip Fractures
Keywords: fragility fractures; hip fractures; augmentation; tip-apex distance
MeSH Terms: conditions — Hip Fractures | interventions — Open Fracture Reduction; Fracture Fixation, Internal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard treatment (Active Comparator): open reduction and internal fixation TFNA
  Interventions: Procedure: open reduction and internal fixation; Device: TFNA
- Augmentation (Experimental): open reduction and internal fixation TFNA Augmentation (Cement)
  Interventions: Procedure: open reduction and internal fixation; Device: TFNA; Device: Augmentation (Cement)

INTERVENTIONS:
Procedure: open reduction and internal fixation — Open reduction and internal fixation using an intramedullary nail
Device: TFNA — Trochanteric Femoral Nail Advance
Device: Augmentation (Cement) — Cement placement (3-6ml) through the cephalic blade under fluoroscopic vision. Cement contains 40% zirconuim dioxide, 15% hydroxiapatite, 45% polymethyl methacrylate (PMMA).
  Arms: Augmentation

SUMMARY:
Randomized clinical trial to assess if the use of augmentation in the treatment of fragility intertrochanteric hip fractures improves radiologic and clinical outcomes in patients aged 65 years or older 1 year after surgery

DETAILED DESCRIPTION:
To determine if the use of augmentation with PMMA in the treatment of fragility intertrochanteric hip fractures improves radiologic and clinical outcomes in osteoporotic patients, investigators aim to conduct a multicentered, randomized, single-blinded clinical trial.

All patients aged 65 years or older arriving to the emergency department of two level-1 trauma centers in Bogotá, Colombia; Hospital Universitario Fundación Santa Fe de Bogotá and Hospital Infantil Universitario de San José, after sustaining a fragility intertrochanteric hip fracture that requires open reduction and internal fixation (ORIF) will be included. These patients must be willing to accept a 1-year follow-up and are required to sign an informed consent agreeing to their participation in the study. For the sample calculation a two-tailed analysis with an alpha-level of significance of 0.05, a power of 80% (β = 0.2) was performed. A total of 35 patients per group plus a 30% increase to control for loss of follow-up was calculated. This gives a total of 90 patients; 45 patients per group.

Patients meeting inclusion and exclusion criteria will be recruited by convenience sampling as they arrive to the emergency department.

Once included in the study, patients will be stratified by age into two groups: patients aged between 65-85 years and patients over 85 years. Then, by using a block randomization, the intervention (augmentation) will be randomly allocated in order to divide the sample population into an intervention group (ORIF + augmentation with PMMA) and a control group (ORIF without augmentation). Randomization will be carried out by the program "Sealed Envelope" (https://www.sealedenvelope.com) that generates a list with codes (each code representing one patient) and randomly assigns them to either the intervention or the control group. This list will be in custody of a research assistant who will not have any contact with patients during the trial's duration and will be in charge of writing the allocation of each code into a sealed, opaque envelope. Each envelope will be given to the surgeon during the procedure at the precise moment where augmentation is needed, revealing whether or not augmentation should be performed. Medical care will be based on Orthogeriatric Programs and surgeries will be performed by orthopaedic surgeons with a clinical fellowship in Orthopaedic Trauma. Patients will be blinded to treatment and will be seen on follow-up visits 15 days, one month, 3 months, 6 months, and 12 months after the procedure.

The primary outcome will be the change in TAD measurement 1 year after the surgical procedure. The functional differences between both groups will be measured as secondary outcomes. Outcomes (primary and secondary) will be measured during follow-up visits one month, 3 months, 6 months, and 12 months after the procedure.

Results will be analyzed using STATA ® Data Analysis and Statistical Software, version 13.1. The sample's demographic and baseline characteristics will be described using descriptive statistics. Continuous variables will be reported as arithmetic means while categorical variables will be reported as absolute values of frequencies and distribution. For the inferential analysis of the results, a Shapiro Wilk W-Test will be used to determine normality distribution of values. If normality assumptions are met, the change in TAD measurement will be analyzed with a student t-test. If not, its non-parametric analogue (Mann-Whitney U-test) will be used. For all other categorical variables, a X2 or Fisher's exact test will be used.

ELIGIBILITY:
Inclusion Criteria:

* patients arriving to the emergency department after sustaining a fragility hip fracture
* radiographic diagnosis of intertrochanteric fracture requiring open reduction and internal fixation
* patient willing to accept a 1-year follow-up
* signature of informed consent

Exclusion Criteria:

* polytrauma
* patients with a non-fragility hip fracture (high-energy trauma)
* hip fractures due to primary or metastatic tumours,
* open or periprosthetic hip fractures
* patients with history of organ transplantation and patients with severe dementia.
* patients with iatrogenic perforation into the hip joint during procedure

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change in TAD measurement | immediate postoperative hip x-ray (starting point), at one month, 3 months, 6 months, and 12 months after the procedure.
  The TAD will be measured in the immediate postoperative hip x-ray, one month, 3 months, 6 months, and 12 months after the procedure.

SECONDARY OUTCOMES:
Parker Mobility Score | one month, 3 months, 6 months, and 12 months after the procedure.
  determine the pre-injury level of mobility and evaluate the functional recovery during the follow-up period.
EQ-5D Questionnaire | one month, 3 months, 6 months, and 12 months after the procedure.
  determine the health-related quality of life perceived by the patient, both before the injury and during the follow-up period
Pain Visual Analogue Scale | one month, 3 months, 6 months, and 12 months after the procedure.
  subjective evaluation of pain intensity

CONTACTS AND LOCATIONS:
Overall Officials: Carlos M Olarte, MD, Principal Investigator — Head of Orthopaedic Department at Hospital Infantil de San José
Locations (2):
- Colombia (2):
  - Fundación Santa Fe de Bogotá, Bogotá, Bogota D.C.
  - Hospital Infantil de San José, Bogotá, Bogota D.C.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kammerlander C, Erhart S, Doshi H, Gosch M, Blauth M. Principles of osteoporotic fracture treatment. Best Pract Res Clin Rheumatol. 2013 Dec;27(6):757-69. doi: 10.1016/j.berh.2014.02.005. PMID 24836334
- [Background] Simunovic N, Devereaux PJ, Sprague S, Guyatt GH, Schemitsch E, Debeer J, Bhandari M. Effect of early surgery after hip fracture on mortality and complications: systematic review and meta-analysis. CMAJ. 2010 Oct 19;182(15):1609-16. doi: 10.1503/cmaj.092220. Epub 2010 Sep 13. PMID 20837683
- [Background] Friedman SM, Mendelson DA, Kates SL, McCann RM. Geriatric co-management of proximal femur fractures: total quality management and protocol-driven care result in better outcomes for a frail patient population. J Am Geriatr Soc. 2008 Jul;56(7):1349-56. doi: 10.1111/j.1532-5415.2008.01770.x. Epub 2008 May 22. PMID 18503520
- [Background] Cooper C, Campion G, Melton LJ 3rd. Hip fractures in the elderly: a world-wide projection. Osteoporos Int. 1992 Nov;2(6):285-9. doi: 10.1007/BF01623184. PMID 1421796
- [Background] Giannoudis PV, Schneider E. Principles of fixation of osteoporotic fractures. J Bone Joint Surg Br. 2006 Oct;88(10):1272-8. doi: 10.1302/0301-620X.88B10.17683. PMID 17012413
- [Background] Moroni A, Larsson S, Hoang Kim A, Gelsomini L, Giannoudis PV. Can we improve fixation and outcomes? Use of bone substitutes. J Orthop Trauma. 2009 Jul;23(6):422-5. doi: 10.1097/BOT.0b013e3181771426. PMID 19550228
- [Background] Kammerlander C, Gebhard F, Meier C, Lenich A, Linhart W, Clasbrummel B, Neubauer-Gartzke T, Garcia-Alonso M, Pavelka T, Blauth M. Standardised cement augmentation of the PFNA using a perforated blade: A new technique and preliminary clinical results. A prospective multicentre trial. Injury. 2011 Dec;42(12):1484-90. doi: 10.1016/j.injury.2011.07.010. Epub 2011 Aug 19. PMID 21855063
- [Background] Kammerlander C, Doshi H, Gebhard F, Scola A, Meier C, Linhart W, Garcia-Alonso M, Nistal J, Blauth M. Long-term results of the augmented PFNA: a prospective multicenter trial. Arch Orthop Trauma Surg. 2014 Mar;134(3):343-9. doi: 10.1007/s00402-013-1902-7. Epub 2013 Dec 3. PMID 24297215
- [Background] Sermon A, Hofmann-Fliri L, Richards RG, Flamaing J, Windolf M. Cement augmentation of hip implants in osteoporotic bone: how much cement is needed and where should it go? J Orthop Res. 2014 Mar;32(3):362-8. doi: 10.1002/jor.22522. Epub 2013 Nov 20. PMID 24259367
- [Background] Eriksson F, Mattsson P, Larsson S. The effect of augmentation with resorbable or conventional bone cement on the holding strength for femoral neck fracture devices. J Orthop Trauma. 2002 May;16(5):302-10. doi: 10.1097/00005131-200205000-00003. PMID 11972072
- [Background] Augat P, Rapp S, Claes L. A modified hip screw incorporating injected cement for the fixation of osteoporotic trochanteric fractures. J Orthop Trauma. 2002 May;16(5):311-6. doi: 10.1097/00005131-200205000-00004. PMID 11972073
- [Background] Mattsson P, Larsson S. Unstable trochanteric fractures augmented with calcium phosphate cement. A prospective randomized study using radiostereometry to measure fracture stability. Scand J Surg. 2004;93(3):223-8. doi: 10.1177/145749690409300310. PMID 15544079
- [Background] Lee PC, Hsieh PH, Chou YC, Wu CC, Chen WJ. Dynamic hip screws for unstable intertrochanteric fractures in elderly patients--encouraging results with a cement augmentation technique. J Trauma. 2010 Apr;68(4):954-64. doi: 10.1097/TA.0b013e3181c995ec. PMID 20386288
- [Background] Dall'Oca C, Maluta T, Moscolo A, Lavini F, Bartolozzi P. Cement augmentation of intertrochanteric fractures stabilised with intramedullary nailing. Injury. 2010 Nov;41(11):1150-5. doi: 10.1016/j.injury.2010.09.026. Epub 2010 Oct 6. PMID 20932521
- [Background] Baumgaertner MR, Solberg BD. Awareness of tip-apex distance reduces failure of fixation of trochanteric fractures of the hip. J Bone Joint Surg Br. 1997 Nov;79(6):969-71. doi: 10.1302/0301-620x.79b6.7949. PMID 9393914
- [Background] Rubio-Avila J, Madden K, Simunovic N, Bhandari M. Tip to apex distance in femoral intertrochanteric fractures: a systematic review. J Orthop Sci. 2013 Jul;18(4):592-8. doi: 10.1007/s00776-013-0402-5. Epub 2013 May 2. PMID 23636573
- [Background] DiMaio FR. The science of bone cement: a historical review. Orthopedics. 2002 Dec;25(12):1399-407; quiz 1408-9. doi: 10.3928/0147-7447-20021201-21. PMID 12502206